CLINICAL TRIAL: NCT05442502
Title: Safety and Efficacy of OGT-assisted Overlap Esophagojejunostomy Versus the Traditional Overlap Method in Laparoscopic Total Gastrectomy for Gastric/Gastroesophageal Junction (G/GEJ) Tumors
Brief Title: Safety and Efficacy of OGT Method Versus the Traditional Overlap Method
Acronym: OGT
Status: Completed | Type: Observational
Sponsor: Nanfang Hospital, Southern Medical University (Other)
Responsible Party: Sponsor
Other Study IDs: NFEC-202204-K17-01
Record Dates: First submitted 2022-06-19; First posted 2022-07-05 (Actual); Last update posted 2022-07-05 (Actual); Status verified 2022-03

CONDITIONS: Gastric Cancer
Keywords: Gastric/gastroesophageal junction (G/GEJ) tumors; Laparoscopy total gastrectomy; Overlap esophagojejunostomy; OGT
MeSH Terms: conditions — Stomach Neoplasms; Neoplasms | interventions — Methods

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- The conventional overlap group: In conventional overlap group, after firing the stapler, two openings were converted into a single entry hole to create an end-to-side esophagojejunostomy, and the entry hole was closed with full-thickness running suture using barbed sutures intracorporeally.
  Interventions: Procedure: The conventional overlap method
- The OGT-assisted group: In OGT group, the anvil fork was inserted into the esophageal mucosa canal by movement of the connection of fork-OGT-gastric tube.
  Interventions: Procedure: The overlap guiding tube(OGT) method

INTERVENTIONS:
Procedure: The overlap guiding tube(OGT) method — The overlap guiding tube(OGT) is used to assist the anvil fork placed into the esophageal cavity.
  Groups: The OGT-assisted group
Procedure: The conventional overlap method — After firing the stapler, two openings were converted into a single entry hole to create an end-to-side esophagojejunostomy, and the entry hole was closed with full-thickness running suture using barbed sutures intracorporeally.
  Groups: The conventional overlap group

SUMMARY:
Introduction: The safety and efficiency of OGT-assisted method have not yet been compared with conventional overlap approach.

Methods Retrospectively analyses the data of 155 gastric/gastroesophageal junction (G/GEJ) cancer patients who underwent laparoscopic total gastrectomy by conventional(conventional group, n=83) or OGT-assisted (OGT group, n=72) overlap methods at Nanfang Hospital. The anastomotic efficiency and surgical outcomes were compared between two groups.

DETAILED DESCRIPTION:
Although our previous multicenter randomized controlled trial (CLASS-01) has confirmed the safety and efficacy of laparoscopic distal gastrectomy for gastric cancer[1, 2], the feasibility of laparoscopic total gastrectomy (LTG) remains uncertain. The most challenging technical difficulty of LTG is esophagojejunostomy(ESJ)[3, 4]. At present, there is still no consensus on the ideal anastomosis method for EJ.

Since overlap esophagojejunostomy was first proposed in 2010[5], it has gradually gone mainstream because of its lower incidence of anastomotic-related complications and satisfactory short-term outcomes[6-10]. However, the overlap approach is technically-difficult and time-consuming, and might confront intraoperative construction complications, such as injuring esophagus caused by the repetition of inserting anvil fork into esophagus or developing esophageal submucosa pseudocanals(video 1 and 2). Therefore, we first designed an overlap guiding tube (OGT)-assisted method to overcame above limitations[11]. And the first reported about the application of OGT-assisted method preliminarily indicated that it is safe and feasible, with a satisfactory success rate of inserting anvil fork into esophageal lumen at first attempt and esophagojejunostomy time[11]. However, the safety and efficiency of OGT-assisted method have not yet been compared side-by-side with the conventional overlap approach. Therefore, this study aimed to compare the OGT-assisted and conventional overlap methods in terms of feasibility and safety in LTG for gastric/gastroesophageal junction (G/GEJ) tumors.

Methods Patients One hundred and fifty-five patients with G/GEJ cancer undergoing LTG via either the conventional overlap esophagojejunostomy(conventional group) or OGT-assisted overlap esophagojejunostomy (OGT group) in the Department of Gastrointestinal Surgery, Southern Medical University Nanfang Hospital, between June 2018 and February 2022 were initially eligible for the study. The inclusion criteria were as follows: (1)gastric cancer was confirmed by pathological examination; (2) tumor located in GEJ with involving esophagus no more than 2cm or the upper, upper to the middle, or entire stomach; (3) had no obvious operative contraindication; and (4) aged 18-85 years. The pathological staging was based on the TNM system of the 8th edition of the International Federation for the prevention and treatment of cancer[12]. This study meets the requirements of the Helsinki Declaration revised in 2013. Patients and their families signed informed consent forms before operation. This study followed the Strengthening the Reporting of Observational Studies in Epidemiology (STROBE) reporting guideline. The data collection protocol was approved by the Ethics Committee of Nanfang Hospital, Southern Medical University. Written informed consent was obtained from all the patients in the study.

ELIGIBILITY:
Inclusion Criteria:

* (1)gastric cancer was confirmed by pathological examination; (2) tumor located in GEJ with involving esophagus no more than 2cm or the upper, upper to the middle, or entire stomach; (3) had no obvious operative contraindication; and (4) aged 18-85 years.

Exclusion Criteria:

* Null.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients enrolled in our study underwent standard LTG with D2 lymphadenectomy according to the Japanese Gastric Cancer Association treatment guidelines
Sampling Method: Non-Probability Sample
Enrollment: 155 (Actual)
Dates: Start 2018-06-01 (Actual); Primary Completion 2022-02-01 (Actual); Study Completion 2022-03-01 (Actual)

PRIMARY OUTCOMES:
The rate of early postoperative complications. | 30 Days
  1. Surgery-related complications: wound complications (infection, effusion, dehiscence,poor healing), intra-abdominal active bleeding,digestive tract active bleeding, anastomotic leakage, anastomotic stenosis, intestinal fistula, pancreatic fistula, chylous fistula, intra-abdominal abscess formation, gastroparesis, intestinal paralysis, intestinal obstruction, cholecystitis, pancreatitis, etc.
  2. System-related complications: pneumonia, pleural effusion, pulmonary embolism, cardiocerebrovascular complications, deep venous thrombosis, urinary tract complications, catheter-related complications, condition of pain,etc.;

SECONDARY OUTCOMES:
The success rate of inserting anvil fork into esophageal lumen at first attempt | 1 Days
  Inserting anvil fork into esophageal lumen at first attempt: when inserting the anvil fork into the esophageal hole, the anvil fork can be correctly placed in a satisfactory position and at a satisfactory angle into the esophageal mucosa canal to be fired for esophagojejunostomy by inserting it only once.
Attempts of inserting anvil fork into esophagus | 1 Days
  The number of times required to try to insert the anvil fork in a satisfactory position and at a satisfactory angle into the esophageal mucosa canal to be fired for esophagojejunostomy.
Time of esophagojejunostomy | 1 Days
  Time of esophagojejunostomy was defined as the time from making the entry hole for the anastomosis on the esophageal stump to the time the common entry hole was closed and reinforced using barbed threads

CONTACTS AND LOCATIONS:
Overall Officials: Jiang Yu, Prof., Principal Investigator — Nanfang Hospital, Southern Medical University
Locations (1):
- Nanfang Hospital, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: Yes
One hundred and fifty-five patients with G/GEJ cancer undergoing LTG via either the conventional overlap esophagojejunostomy(conventional group) or OGT-assisted overlap esophagojejunostomy (OGT group) in the Department of Gastrointestinal Surgery, Southern Medical University Nanfang Hospital, between June 2018 and February 2022 were initially eligible for the study. The inclusion criteria were as follows: (1)gastric cancer was confirmed by pathological examination; (2) tumor located in GEJ with involving esophagus no more than 2cm or the upper, upper to the middle, or entire stomach; (3) had no obvious operative contraindication; and (4) aged 18-85 years.
Supporting Information: Study Protocol
Time Frame: July,2022-December 2023.
Access Criteria: All accessing are approved.